CLINICAL TRIAL: NCT00916461
Title: A Randomised, Double Blind Pilot Study of Minocycline and Placebo Added to Treatment-as-Usual (TAU) in First-Episode Psychosis
Brief Title: Role of Minocycline in First Episode Psychosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanley Medical Research Institute (Other)
Collaborators: Institute of Psychiatry, Rawalpindi Medical College, Pakistan (Unknown); Pakistan Institute of Living and Learning (Other); University of Sao Paulo (Other)
Responsible Party: Dr Imran B Chaudhry, University of Manchester
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: SMRI 04T-583
Record Dates: First submitted 2009-06-08; First posted 2009-06-09 (Estimated); Last update posted 2009-06-15 (Estimated); Status verified 2009-06

CONDITIONS: First Episode Psychosis
Keywords: First episode psychosis; Schizophrenia; Minocycline; neuroprotection; First episode non affective psychosis; With in first five years of illness
MeSH Terms: conditions — Schizophrenia; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minocycline (Active Comparator)
  Interventions: Drug: Minocycline
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minocycline — Minocycline + treatment as usual. 50 mg twice daily increasing to 200 mgs per day, increments of 50 mgs every 2 weeks.
  Arms: Minocycline
Drug: Placebo — Placebo + treatment as usual.
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to determine whether the addition of minocycline or placebo to treatment as usual (TAU):

1. prevents the accumulation of negative symptoms and intellectual decline following a first episode of non-affective psychosis; and
2. whether minocycline stabilizes the efficacy of antipsychotics.

DETAILED DESCRIPTION:
Background:

There is increasing clinical, neuropsychological and imaging evidence that schizophrenia involves a progressive process at the time of the first episode and later in life. However, it is not clear which systems are affected nor in which parts of the brain. In two Stanley first episode cohorts at Manchester (Stirling et al, 2004,) and in a group of elderly patients with schizophrenia (Gabrovska-Johnson et al 2004), evidence of deterioration in visuo-spatial functions has been found. This implies a right-hemisphere pathology. Other evidence suggests that the initiation of schizophrenia may involve left-sided pathology (Lawrie et al 2002) so it could be that right hemisphere pathology may follow left and give rise to the deficits of chronic schizophrenia (Gabrovska-Johnson et al 2004). If so, early treatment with a neuroprotective agent might prevent the accumulation of deficit symptoms and cognitive impairment.

Minocycline is a tetracycline antibiotic with proven long-term high dose safety in humans, is routinely used to treat acne and rheumatoid arthritis demonstrating that it acts as a non-steroidal anti-inflammatory, as well as an antimicrobial drug. Minocycline, unlike tetracycline, crosses the blood-brain barrier. This and related compounds show neuroprotective properties in rat models of ischemic brain damage, in glutamate neurotoxicity in cell cultures and in a rat model of Huntington's disease in which it slowed progression (Chen et al, 2000; Yrjanheikki et al, 1999). Minocycline delays disease onset and extends survival in amyotrophic lateral sclerotic mice (Shan Zhu et al 2002).

Minocycline has various properties including inhibition of capsases, inhibition of microglial activation, reduced cyclooxygenase-2 expression and reduced prostaglandin E (2) formation. Furthermore, it inhibits the formation of inducible nitric oxide - a mechanism of glial activation. All these mechanisms have been implicated in schizophrenia. All these mechanisms have been implicated in schizophrenia.

Because of its broad spectrum of action, we consider minocycline is an important candidate molecule for the prevention of deterioration in schizophrenia. Based on the evidence so far we propose a randomised double blind placebo controlled study of minocycline added to treatment-as-usual (TAU) in first-episode psychosis.

Study Hypotheses:

* A neurodegenerative process, initially most marked in the left hemisphere, in late adolescence is responsible for the onset of schizophrenia in those at risk.
* Continuation of this process after onset and its extension to the right hemisphere causes accumulation of deficit symptoms and cognitive decline.
* Glutamate antagonism may enhance the antipsychotic effects of dopamine receptor blockade and prevent attenuation of efficacy with long-term treatment.

TREATMENT:

Minocycline is a widely available antibiotic given in doses of 50mg twice daily increasing to 200mgs per day. It has been used very widely and appears to be tolerated well. The study advisor, Dr. Serdar Dursun, has used doses of up to 200mg per day in the treatment of Huntington's disease (Denovan-Wright et al 2002).

It is widely available in Pakistan and Brazil and given in doses of 50mg twice daily increasing to 100mg twice daily (in total 200mg per day) (British National Formulary: BNF maximum dose 200mg per day). As per counselling recommendations in the British National Formulary: "minocycline medication should be swallowed whole with plenty of fluid while sitting or standing", to allow effective absorption. Patients will be counselled that 'the study medication should be swallowed whole with plenty of fluid while standing or sitting.'

Patients will be informed regarding reported side-effects as cited in the BNF these include; nausea, vomiting, diarrhoea, dysphagia, oesophageal irritation, anorexia, dizziness, tinnitus, vertigo, hypersensitivity reactions (rash, exfoliative dermatitis, urticaria, angioedema, anaphylaxis, pericarditis), headache, visual disturbances, hepatotoxicity, pancreatitis, antibiotic associated colitis, blood dyscrasias, exacerbation of systemic lupus erythematosus and myasthenia gravis, rarely photosensitivity, skin, teeth, conjunctiva, tears and sweat discoloration.

NUMBER OF PATIENTS:

Using data from the SOCRATES study, we are able to calculate that 40 patients per treatment arm will detect a group difference on the primary outcome measure, i.e, PANSS, giving a 85% chance of detecting a difference between treatment groups of 4 points. The power estimate is likely to be conservative as there are three treatment groups. The automated CSF measures will detect a 5% group difference with these sample sizes. A minimum of 52 completed patients will be necessary (26 completed patients per treatment group).

Study Advisors:

Prof Bill Deakin(design), Prof Serdar Dursun(scientific), Prof Shon Lewis (clinical), Dr John Stirling (cognition), Dr Paul Richardson (cognition), Prof Graham Dunn (analysis).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* Diagnostic and Statistical Manual-IV (DSM-IV) diagnosed first episode psychosis, schizophrenia, schizoaffective disorder, psychosis not otherwise specified or schizophreniform disorder
* First episode (within first 5 years of diagnosis)
* Competent and willing to give informed consent
* Medication remained stable 4 weeks prior to baseline
* Able to take oral medication and likely to complete the required evaluations
* Female participants of child bearing capability must be willing to use adequate contraceptives for the duration of the study, and, willing to have a pregnancy test pre-treatment and at ten weekly intervals while on study medication

Exclusion Criteria:

* Relevant medical illness [renal, hepatic, cardiac, serious dermatological disorders such as exfoliative dermatitis, systemic lupus erythematosus (SLE)] in the opinion of the investigators (see section 6.2a)
* Prior history of intolerance to any of the tetracyclines
* Concomitant penicillin therapy
* Concomitant anticoagulant therapy
* Presence of a seizure disorder, not including clozapine-induced seizures
* Presently taking valproic acid
* Any change of psychotropic medications within the previous six weeks
* Diagnosis of substance abuse (except nicotine or caffeine) or dependence within the last three months according to DSM-IV criteria
* Pregnant or breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Positive and negative symptoms on Positive and Negative Syndrome Scale (PANSS) | Baseline and 12 months

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) | Baseline and 12 months
Global Assessment of Functioning (GAF) | Baseline and 12 months
Abnormal Involuntary Movement Scale (AIMS) | Baseline and 12 months
Assessment of side effects | Baseline and 12 months
Doses of antipsychotic drugs | Baseline and 12 months
neurocognitive test scores | Baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Imran B Chaudhry, MD, Principal Investigator — University of Manchester; Jaime EC Hallak, MD, Study Director — University of San Paulo, Brazil; Nusrat Husain, MD, Study Director — University of Manchester
Locations (4):
- Department of Neurology, Psychiatry and Psychological Medicine, University of San Paulo, São Paulo, Brazil
- Pakistan (3):
  - Civil Hospital Karachi, Karachi
  - Karwan e Hayat, Karachi
  - Institute of Psychiatry, Rawalpindi medical College, Rawalpindi

REFERENCES:
- [Background] Chen M, Ona VO, Li M, Ferrante RJ, Fink KB, Zhu S, Bian J, Guo L, Farrell LA, Hersch SM, Hobbs W, Vonsattel JP, Cha JH, Friedlander RM. Minocycline inhibits caspase-1 and caspase-3 expression and delays mortality in a transgenic mouse model of Huntington disease. Nat Med. 2000 Jul;6(7):797-801. doi: 10.1038/77528. PMID 10888929
- [Background] Gabrovska-Johnson VS, Scott M, Jeffries S, Thacker N, Baldwin RC, Burns A, Lewis SW, Deakin JF. Right-hemisphere encephalopathy in elderly subjects with schizophrenia: evidence from neuropsychological and brain imaging studies. Psychopharmacology (Berl). 2003 Sep;169(3-4):367-75. doi: 10.1007/s00213-003-1524-9. Epub 2003 Jul 4. PMID 12845412
- [Background] Yrjanheikki J, Tikka T, Keinanen R, Goldsteins G, Chan PH, Koistinaho J. A tetracycline derivative, minocycline, reduces inflammation and protects against focal cerebral ischemia with a wide therapeutic window. Proc Natl Acad Sci U S A. 1999 Nov 9;96(23):13496-500. doi: 10.1073/pnas.96.23.13496. PMID 10557349
- [Background] Stirling J, White C, Lewis S, Hopkins R, Tantam D, Huddy A, Montague L. Neurocognitive function and outcome in first-episode schizophrenia: a 10-year follow-up of an epidemiological cohort. Schizophr Res. 2003 Dec 15;65(2-3):75-86. doi: 10.1016/s0920-9964(03)00014-8. PMID 14630300
- [Background] Zhu S, Stavrovskaya IG, Drozda M, Kim BY, Ona V, Li M, Sarang S, Liu AS, Hartley DM, Wu DC, Gullans S, Ferrante RJ, Przedborski S, Kristal BS, Friedlander RM. Minocycline inhibits cytochrome c release and delays progression of amyotrophic lateral sclerosis in mice. Nature. 2002 May 2;417(6884):74-8. doi: 10.1038/417074a. PMID 11986668
- [Background] Denovan-Wright EM, Devarajan S, Dursun SM, Robertson HA. Maintained improvement with minocycline of a patient with advanced Huntington's disease. J Psychopharmacol. 2002 Dec;16(4):393-4. doi: 10.1177/026988110201600417. PMID 12503842